CLINICAL TRIAL: NCT02297061
Title: Study on the Value of Thrombelastogralhy to Pre-operatively Predict Hip Fracture Patients at Risk of Major Blood Loss During and After Surgery.
Brief Title: Can Thrombelastography Predict Blood Loss in Patients With Hip Fractures
Status: Completed | Type: Observational
Sponsor: Hvidovre University Hospital (Other)
Collaborators: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Peter Toft Tengberg, Principal investigator, Hvidovre University Hospital
Other Study IDs: TEGHIP
Record Dates: First submitted 2014-02-09; First posted 2014-11-21 (Estimated); Last update posted 2014-11-21 (Estimated); Status verified 2014-11

CONDITIONS: Hip Fracture; Blood Loss
Keywords: Hip fracture; Thrombelastography; Blood loss
MeSH Terms: conditions — Hip Fractures; Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- TEG group: 200 consecutive hip fracture patients, Thrombelastography is performed on admission.
  Interventions: Biological: Thrombelastography analysis (TEG)

INTERVENTIONS:
Biological: Thrombelastography analysis (TEG) — TEG analysis is performed on admission

SUMMARY:
Hip fractures are associated with a large hidden blood loss. That is, the total blood loss associated with hip fracture surgery is much greater than that observed intra operatively. There is currently no viable method of identifying patients at risk of transfusion. The on admission haemoglobin level has been shown to be falsely reassuring .

We are conducting a study of 200 consecutive hip fracture patients. Thrombelastography (TEG) is taken on admission. The results are blinded to clinicians. Results will be evaluated at the end of the study, comparing intra-operative and total blood losses with the TEG profile of the patient.

DETAILED DESCRIPTION:
Hip fractures are associated with a large hidden blood loss. That is, the total blood loss associated with hip fracture surgery is much greater than that observed intra operatively. The total blood loss depends on the type of fracture and associated surgery. Extra-capsular fractures treated with an intramedullary nail are thus associated with the largest hidden blood loss with a median of approximately 1500 ml . This hidden blood loss is primarily associated with the trauma and fracture itself and not, as such, with the surgical procedure.

Postoperative anaemia necessitating transfusion and a haemoglobin level below 8 g per dL, in hip fracture patients, are both associated with an increased mortality Controversy remains on the benefits and indications for transfusion in this group of patients.

There is currently no viable method of identifying patients at risk of transfusion. The on admission haemoglobin level has been shown to be falsely reassuring . TEG has to our knowledge only been used in one previous study of hip fractures. The outcome measure in this study was thromboembolic events. We have not been able to identify any studies on the use of TEG, INR, APTT or other tests as predictors of blood loss in hip fracture patients.

Clinicians would greatly benefit from a tool to predict the at-risk patient on admission. TEG has been suggested as such a tool. Bolliger et al suggests that TEG can be used in goal-oriented algorithms to optimize targeted transfusion therapies in trauma patients or patients undergoing major surgery. We hypothesize that TEG can be used for this purpose in patients with hip fracture. These patients can have large blood losses and they sustain the double trauma of a hip fracture and major orthopaedic surgery.

ELIGIBILITY:
Inclusion Criteria:

* All hip fracture patients admitted through the emergency room (ER) at Hvidovre University Hospital in the study period.

Exclusion Criteria:

* Hip fracture patients who are transfered from other wards in the hospital do not go through the ER and are not included.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Hip fracture patients admitted to Hvidovre University Hospital in the study period.
Sampling Method: Probability Sample
Enrollment: 180 (Actual)
Dates: Start 2013-12; Primary Completion 2014-05 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Total blood loss compared to TEG profile on admission | 4 days postoperatively
  TEG profiles will be compared to the blood losses of the patients, after completion of the study.

SECONDARY OUTCOMES:
Thrombotic incidences | 90 days after operation
  Can TEG analysis predict thrombotic incidences in hip fracture patients.
Mortality | 90 days after operation
  Relation between TEG values and mortality.

CONTACTS AND LOCATIONS:
Overall Officials: Peter T Tengberg, MD, Principal Investigator — Hvidovre University Hospital
Locations (1):
- Hvidovre University Hospital, Hvidovre, Denmark